CLINICAL TRIAL: NCT07148115
Title: Pregnancy Outcomes Prior to a Systemic Lupus Erythematosus Diagnosis
Brief Title: Pregnancies Before the Diagnosis of Systemic Lupus Erythematosus
Acronym: PREDILUP
Status: Recruiting | Type: Observational
Sponsor: University of Algiers (Other)
Responsible Party: Principal Investigator, W.N. Nibouche-Hattab, Professor of Medicine, University of Algiers
Other Study IDs: LES/PRG/24
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-08

CONDITIONS: Pregnancy Complications; SLE
Keywords: Pregnancy; SLE; Obstetrical events
MeSH Terms: conditions — Pregnancy Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Femelle patients at procreation age with diagnosis of LES: Patients that have had pregnancies history before the diagnosis of LES
  Interventions: Other: Collect data on all pregnancies before and after diagnosis of SLE.

INTERVENTIONS:
Other: Collect data on all pregnancies before and after diagnosis of SLE. — For participants who are still alive, data are collected from interviews with patients using a prepared questionnaire that asks about all pregnancies and obstetrical events prior to the diagnosis of SLE.
  For deceased patients, data are taken from the medical records of obstetrical events.
  Data will be collected on anthropometric, biological, immunological, and histological features before and after the diagnosis of SLE, if available.
  The activity and severity of the disease after diagnosis will be assessed using the recommended tools.

SUMMARY:
This is an observational, monocentric, retrospective cohort study. Its primary objective is to examine maternal and foetal outcomes in pregnancies that occurred before the diagnosis of systemic lupus erythematosus (SLE) in a group of female participants who were subsequently diagnosed with the condition.

DETAILED DESCRIPTION:
The investigators aim to study obstetrical and systemic signs in participants' pregnancies prior to an SLE diagnosis. Information will be collected from medical records and by asking participants questions during medical visits. The diagnosis of SLE is made using the ACR 1997 criteria. It is also based on renal histological findings.

The study must answer three questions:

1. Are systemic signs of SLE present before or during pregnancy?
2. What were the fetal and maternal outcomes after or during each pregnancy? What is/was the severity of SLE after diagnosis?

ELIGIBILITY:
Inclusion criteria:

* Women of childbearing age with a history of at least one pregnancy
* Pregnancy occurred before the diagnosis of LES.
* LES was diagnosed after at least one pregnancy.
* The subject is classified as having LES according to the 1997 ACR or EULAR 2019 criteria.

Exclusion criteria:

LES was previously diagnosed prior to any conception.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only biological femelle sex and cis-gender people that have experienced pregnancy are eligible to participate to the study
Study Population: Eligible patients for the study are selected from all women diagnosed with lupus erythematosus in the Department of Internal Medicine at the Ain-Taya Teaching Hospital from 2000 to 2025. Patients are recruited from primary care, emergency units, or the gynecology and obstetrics department. These patients are being followed up in the Department of Internal Medicine at Ain-Taya Hospital.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
1. Primary outcome: Prevalence of obstetrical events before the diagnosis of SLE. Secondary outcome: 1. Assess the severity of the disease at the time of LES diagnosis. 2. Compare the outcomes of pregnancies before and after the LES | The patient will be assessed from the beginning of each pregnancy and in the three month after childbirth
  * Evaluate the number of pregnancies for each woman before and after the diagnosis of lupus.
  * Assess obstetric events for each pregnancy (spontaneous abortion, prematurity, fetal death, pre-eclampsia, HELLP syndrome, or other pregnancy-related events).
  * Assess the presence of systemic signs during pregnancy or the postpartum period.
  * Collect data on the baby's status, including weight, height, and any morbid conditions (dermatological, cardiac, respiratory, etc.).
  * Note the timeframe between the last pregnancy or delivery and the SLE diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Wafia-Nadia Nibouche-Hattab, Professor of medicine, Study Director — University of Algiers. Faculty of medicine
Locations (2):
- Algeria (2):
  - Department of internal medicine, Ain-Taya's teaching Public hospital, Aïn Taya, Algiers Province
  - Ain-Taya's Public Hospital, Algiers

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One month after the end of the study, presumely in March 2026 until Avril 2026
Access Criteria: the reviewers board of journal if manuscript is accepted. they will be able to access all data collected and statistical study.
URL: https://drive.google.com/drive/my-drive